CLINICAL TRIAL: NCT06713005
Title: The Clinical Efficacy of Different Durations of Suprascapular Nerve Pulsed Radiofrequency Treatment in Chronic Soulder Pain
Brief Title: The Clinical Efficacy of Different Durations of Suprascapular Nerve Pulsed Radiofrequency
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hanzade Aybuke Unal, Principal Investigator, Ankara University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/765
Record Dates: First submitted 2024-11-26; First posted 2024-12-03 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Suprascapular Nerve; Shoulder Impingement Syndrome; Pulsed Radiofrequency; Chronic Pain; Supraspinatus Tendinopathy
Keywords: pulsed radiofrequency; suprascapular nerve; chronic pain; impingement syndrome; Supraspinatus tendinopathy
MeSH Terms: conditions — Shoulder Impingement Syndrome; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Group 1: 4 mins suprascapular pulsed RF Group 2: 9 mins suprascapular pulsed RF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4 min suprascapular pulsed RF (Other): Suprascapular nerve pulsed RF is applied for 4 minutes.
  Interventions: Procedure: suprascapular nerve block and 4 mins Pulsed radiofreuency application to suprascapular nerve
- 9 min suprascapular pulsed RF (Other): Suprascapular nerve pulsed RF is applied for 8 minutes.
  Interventions: Procedure: suprascapular nerve block and 9 mins Pulsed radiofreuency application to suprascapular nerve

INTERVENTIONS:
Procedure: suprascapular nerve block and 4 mins Pulsed radiofreuency application to suprascapular nerve — suprascapular nerve pulsed rf
  Arms: 4 min suprascapular pulsed RF
Procedure: suprascapular nerve block and 9 mins Pulsed radiofreuency application to suprascapular nerve — suprascapular nerve block and 4 mins Pulsed radiofreuency application to suprascapular nerve
  Arms: 9 min suprascapular pulsed RF

SUMMARY:
Chronic shoulder pain due to impingement syndrome and supraspinatus tendinosis is a debilitating condition. Suprascapular nerve innervates most part of shoulder joint. Supraspinatus nerve block can be used as a part of pain therapy. However, its efficacy is short-lasting. To prolong analgesia, short bursts of electrical stimulation to suprascapular nerve may be applied. To the date there is no consensus about duration of these type of stimulation. Investigators' aim is to investigate efficacy of two different duration of stimulation (pulsed radiofrequency) on chronic shoulder pain.

DETAILED DESCRIPTION:
Pulsed radiofrequency (pRF) treatment of suprascapular nerve can be used successfully to alleviate pain due to shoulder impingement syndrome and supraspinatus tendinosis. Radiofrequency waves produced by radiofrequency (RF) generator through pRF modality are applied to suprascapular nerve and create magnetic field. This field leads to pain modulation by changing neuronal activity and resulting in long term depression of pain transmitting nerve fibers. Temperature around nerve never exceeds 42 degree and by this way the nerve can be protected from coagulation necrosis and demiyelinisation. pRF can be used in the treatment of mixed type nerves such as suprascapular nerve. There are preclinical and clinical studies which report that with longer pRF duration, more favorable analgesia. Suprascapular pRF is performed with 22G, 10 cm, 5 mm active lead RF needle via USG guided posterior approach as institution procotol. Howeveri clinicians can choose any duration of pRF. Instution's pain medicine practitioners HAU and GEO choose 4 and 9 minutes of pRF duration, respectively. Investigators' aim is to investigate the efficacy of two different pRF duration, 4 and 9 minutes, on Shoulder Pain and Disability Index (SPADI) and Numeric Rating Scale-11(NRS-11) at 3 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years
* Shoulder pain caused by impingement syndrome
* Shoulder pain due to supraspinatus tendinosis
* Diagnosis of impingement syndrome and supraspinatus tendinosis confirmed through physical examination and radiological imaging (MRI)
* Pain persisting for 3 months or longer
* Numeric Pain Rating Scale (NRS) score of 4 or higher despite conservative treatment

Exclusion Criteria:

* Patients unwilling to participate in the study
* Presence of chronic pain due to other conditions
* Presence of cervical radiculopathy
* History of opioid use
* Uncontrolled diabetes (HbA1c > 8)
* History of shoulder surgery on the affected side
* Uncontrolled psychiatric disorders despite medical treatment
* History of cancer
* History of stroke

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Postprocedure 3th month pain severity | From procedure to 3 months after prodecure
  Severity of pain will be assessed with Numeric Rating Scale (NRS-11) at baseline, 1 weeks, 1 months and 3 months after interventions. NRS-11 is a 11 point likert type scale. Higher scores represent more severe pain.

SECONDARY OUTCOMES:
Postprocedure pain severity at first week | From procedure to 1 week after procedure
  Severity of pain will be assessed with Numeric Rating Scale (NRS-11) at 1 week after interventions. NRS-11 is a 11 point likert type scale. Higher scores represent more severe pain.
Postprocedure first month pain severity | From procedure to 1 month after procedure
  Severity of pain will be assessed with Numeric Rating Scale (NRS-11) at 1 month after interventions. NRS-11 is a 11 point likert type scale. Higher scores represent more severe pain.
Postprocedure SPADI scores at first week | From procedure to 1 week after procedure
  Functionality will be assessed with Shoulder Pain and Disability Index (SPADI) at 1 week. SPADI measures pain and disability related shoulder function. SPADI has 0 minimum and 100 maximum value. Lower scores represent better outcomes.
Postprocedure first month SPADI scores | From procedure to 1 month after procedure
  Functionality will be assessed with Shoulder Pain and Disability Index (SPADI) at 1 month. SPADI measures pain and disability related shoulder function. SPADI has 0 minimum and 100 maximum value. Lower scores represent better outcomes.
Postprocedure 3th month SPADI scores | From procedure to 3 month after procedure
  Functionality will be assessed with Shoulder Pain and Disability Index (SPADI) at 3th month. SPADI measures pain and disability related shoulder function. SPADI has 0 minimum and 100 maximum value. Lower scores represent better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Güngör Enver Özgencil, Prof Dr, Study Director — Ankara University School of Medicine Department of Anesthesiology and Reanimation
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All data can be shared except personal data.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 5 years after January 2026
Access Criteria: Upon reasonable request

REFERENCES:
- [Background] Gupta SK, Ghai B, Makkar JK, Dhiman D, Chouhan DK. Effectiveness of ultrasound-guided pulsed radiofrequency ablation of suprascapular nerve versus local anaesthetics with steroids in patients with chronic shoulder pain: A randomised controlled trial. Indian J Anaesth. 2024 Aug;68(8):731-734. doi: 10.4103/ija.ija_939_23. Epub 2024 Jul 2. No abstract available. PMID 39176114